CLINICAL TRIAL: NCT06280924
Title: Multiple Myeloma Exercise Prehabilitation for Individuals Awaiting a Stem Cell Transplantation (MOTIVATE): A Randomized Controlled Feasibility Trial
Brief Title: Prehab Prior to Stem Cell Transplantation in Multiple Myeloma
Acronym: MOTIVATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HREBA.CC-23-0220
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Multiple Myeloma; Exercise; Prehabilitation
MeSH Terms: conditions — Multiple Myeloma; Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: An independent assessor will conduct the post-intervention assessment. The independent assessor will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator): Participants in this group will receive exercise counseling as per standard care for 10-weeks. This will include: (1) counseling on remaining active during chemotherapy; (2) handouts on the benefits of exercise during chemotherapy, exercise behavior change strategies, and how to exercise safely. Participants will be encouraged to remain as physical active as possible. As per American College of Sports Medicine 2019 guidelines, participants will be advised to take part in moderate intensity exercise for a total of 90 minutes per week.
  Interventions: Behavioral: Standard Care
- Supported Exercise Group (Experimental): Participants assigned to the exercise group will take part in a 10-week exercise program delivered in-person and through the HEAL-ME app. The program comprises (1) a minimum of one supervised session (in-person or virtual through a Zoom platform embedded in HEAL-ME), (2) a minimum of one independent exercise workout within the HEAL-ME app, and (3) exercise specific education content as per standard care.
  Interventions: Behavioral: Supported Exercise

INTERVENTIONS:
Behavioral: Supported Exercise — Participants will take part in a prehabilitation exercise program prior to undergoing a stem cell transplant.
  Arms: Supported Exercise Group
Behavioral: Standard Care — Participants will receive standard care
  Arms: Standard Care

SUMMARY:
The primary purpose of this study is to see if individuals with Multiple Myeloma are able and interested in taking part in a tailored exercise program while undergoing their chemotherapy prior to a stem cell transplant. We also hope to learn if this type of program, along with a flexible delivery format (in-person and virtual), helps in maintaining or improving physical fitness, muscle mass and strength, and quality of life during chemotherapy.

DETAILED DESCRIPTION:
MOTIVATE is a multi-methods feasibility randomized trial. We will recruit a minimum of 30 individuals with multiple myeloma who are undergoing chemotherapy prior to a Stem Cell Transplant. The study will be conducted in two phases:

Phase I: Feasibility Study The aim of this phase is to determine the feasibility and preliminary effectiveness of a 10-week exercise intervention compared to physical activity counseling alone.

Phase II: Qualitative Study The aim of this phase is to evaluate the acceptability of the Healthy Eating Active Living (HEAL-ME) app design, program delivery/design, and perceived effectiveness of the intervention at the level of the participant.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of Multiple Myeloma
2. Be transplant eligible
3. Be undergoing chemotherapy prior to, or following an autologous stem cell transplant as part of their cancer treatment; or transplant ineligible.
4. Be an Alberta resident
5. Be ≥18 years of age
6. Be able to read and understand English.

Exclusion Criteria:

1. Their disease status/comorbidities preclude exercise testing or participation
2. They are unable to commit to the 10-week exercise program and/or testing sessions at the Cancer Rehabilitation Clinic at the University of Alberta
3. They do not have regular access to the internet and/or an electronic device in the home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Study completion rate | 10-weeks
  The percentage of participants who complete the study, including the intervention and follow-up assessment

SECONDARY OUTCOMES:
Recruitment rate | 18 months
  The percentage of participants who are eligible and consent to participate in the study.
Attendance rate | 18 months
  The percentage of group and individual exercise sessions completed over the 10 weeks.
Edmonton Symptom Assessment System | 10 weeks
  Tool to assess 11 symptoms related to cancer: higher scores reflect worse symptom burden
Functional Assessment of Cancer Therapy Multiple Myeloma | 10 weeks
  Health-related quality of life questionnaire: higher scores reflect better quality of life
Functional Assessment of Cancer Therapy: Fatigue Subscale (13-item) | 10 weeks
  Fatigue questionnaire: higher scores reflect less fatigue
Body weight | 10 weeks
  Weight measured in kilograms
Body height | 10 weeks
  Weight measured in centimetres (to nearest 0.5 cm)
Grip Strength | 10 weeks
  Hand grip measured in kilograms using a dynamometer
Calf muscle size | 10 weeks
  Calf circumference measured in centimetres to the nearest 0.1 cm
Thigh muscle thickness | 10 weeks
  Ultrasound measurement of rectus femoris muscle cross-sectional area
Short Physical Performance Battery | 10 weeks
  Test includes 4-meter timed walk, balance and 5-repetition sit-to-stand
Six-minute walk test | 10 weeks
  Distance covered in metres (to nearest cm) in 6 minutes (hallway)
One leg stance balance | 10 weeks
  Time standing on one foot (to a maximum of 45 seconds)
Shoulder flexion range of motion | 10 weeks
  Upper limb flexibility measured in degrees
Sit and reach test | 10 weeks
  Lower limb flexibility measured in cms (to nearest 0.5 cm)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Sellar, PhD, Study Director — University of Alberta
Locations (1):
- University of Alberta/ Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data generated or analyzed during this study will be available in the University of Alberta Dataserve repository
Supporting Information: Study Protocol, SAP
Time Frame: Data will be deposited approximately one-year after completion of the study
Access Criteria: Open access